CLINICAL TRIAL: NCT02415439
Title: A Phase 1 Randomized, Placebo-Controlled, Double-Blind, Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of VBP15 in Healthy Adult Subjects
Brief Title: A Phase 1 Single Ascending Dose and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of VBP15 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ReveraGen BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VBP15-001
Record Dates: First submitted 2015-03-02; First posted 2015-04-14 (Estimated); Results first posted 2017-01-05 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Safety; tolerability; pharmacokinetics; adult; volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (13):
- VBP15- 0.1 mg/kg SAD (Experimental): Subjects were orally administered a single dose of VBP15 at 0.1 mg/kg under fasted conditions.
  Interventions: Drug: VBP15
- VBP15- 0.3 mg/kg SAD (Experimental): Subjects were orally administered a single dose of VBP15 at 0.3 mg/kg under fasted conditions.
  Interventions: Drug: VBP15
- VBP15- 1.0 mg/kg SAD (Experimental): Subjects were orally administered a single dose of VBP15 at 1.0 mg/kg under fasted conditions.
  Interventions: Drug: VBP15
- VBP15- 3.0 mg/kg SAD (Experimental): Subjects were orally administered a single dose of VBP15 at 3.0 mg/kg under fasted conditions.
  Interventions: Drug: VBP15
- VBP15- 8.0 mg/kg Fasting SAD (Experimental): Subjects were orally administered a single dose of VBP15 at 8.0 mg/kg under fasted conditions.
  Interventions: Drug: VBP15
- VBP15- 8.0 mg/kg Fed SAD (Experimental): Subjects were orally administered a single dose of VBP15 at 8.0 mg/kg within 30 minutes of beginning a high fat/high high calorie meal.
  Interventions: Drug: VBP15
- VBP15- 20.0 mg/kg SAD (Experimental): Subjects were orally administered a single dose of VBP15 at 20.0 mg/kg under fasted conditions.
  Interventions: Drug: VBP15
- Placebo - SAD (Placebo Comparator): Subjects were orally administered a placebo under fasted conditions.
  Interventions: Drug: Placebo
- VBP15- 1.0 mg/kg 14 Day MAD (Experimental): Subjects were orally administered VBP15 at 1.0 mg/kg for 14 days under fasted conditions.
  Interventions: Drug: VBP15
- VBP15- 3.0 mg/kg 14 Day MAD (Experimental): Subjects were orally administered VBP15 at 3.0 mg/kg for 14 days under fasted conditions.
  Interventions: Drug: VBP15
- VBP15- 9.0 mg/kg 14 Day MAD (Experimental): Subjects were orally administered VBP15 at 9.0 mg/kg for 14 days under fasted conditions.
  Interventions: Drug: VBP15
- VBP15- 20.0 mg/kg 14 Day MAD (Experimental): Subjects were orally administered VBP15 at 20.0 mg/kg for 14 days under fasted conditions.
  Interventions: Drug: VBP15
- Placebo MAD (Placebo Comparator): Subjects were orally administered placebo for 14 days under fasted conditions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VBP15
  Arms: VBP15- 0.1 mg/kg SAD; VBP15- 0.3 mg/kg SAD; VBP15- 1.0 mg/kg 14 Day MAD; VBP15- 1.0 mg/kg SAD; VBP15- 20.0 mg/kg 14 Day MAD; VBP15- 20.0 mg/kg SAD; VBP15- 3.0 mg/kg 14 Day MAD; VBP15- 3.0 mg/kg SAD; VBP15- 8.0 mg/kg Fasting SAD; VBP15- 8.0 mg/kg Fed SAD; VBP15- 9.0 mg/kg 14 Day MAD
Drug: Placebo
  Arms: Placebo - SAD; Placebo MAD

SUMMARY:
The purpose of this study is to examine the safety, tolerability, and PK of various increasing single and multiple doses of VBP15 in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* For the Single Ascending Dose Study (SAD): Male subjects, ages 18 to 65 years, inclusive.
* For the Multiple Ascending Dose Study (MAD): Male subjects or female subjects of nonchildbearing potential ages 18 to 65, inclusive.

Exclusion Criteria:

* For the MAD Study: Women of childbearing potential.
* Clinically significant abnormal laboratory parameters

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2015-01; Primary Completion 2015-11 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PRA Health Sciences, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In the single ascending dose (SAD) study, subjects were assigned to 1 of 7 dose groups and received a single oral dose of VBP15 or placebo. The multiple ascending dose (MAD) was initiated after a review of safety data from SAD groups. In the MAD study, subjects were randomized to 1 of 4 groups to receive VBP15 or placebo once daily for 14 days
Pre-assignment Details: An escalating-dose design was chosen for the SAD and MAD studies to allow increase of the dose after assessment of safety and tolerability of each preceding dose. Escalation to the next higher dose was performed using a factor of 3 for each subsequent dose until a maximum of 20 mg/kg was reached. No subject received more than 1 dose level of VBP15.
Groups:
- VBP15- 8.0 mg/kg Fasted SAD: Subjects were orally administered a single dose of VBP15 at 8.0 mg/kg under fasted conditions.
- VBP15- 8.0 mg/kg Fed SAD: Subjects were orally administered a single dose of VBP15 at 8.0 mg/kg within 30 minutes of beginning a high fat/high calorie meal.
- Placebo SAD: Subjects were orally administered a single dose of placebo under fasted conditions.
- VBP15- 1.0 mg/kg 14 Day MAD: Subjects were orally administered VBP15 at 1.0 mg/kg daily for 14 days under fasted conditions.
- VBP15- 3.0 mg/kg 14 Day MAD: Subjects were orally administered VBP15 at 3.0 mg/kg daily for 14 days under fasted conditions.
- VBP15- 9.0 mg/kg 14 Day MAD: Subjects were orally administered VBP15 at 9.0 mg/kg daily for 14 days under fasted conditions.
- VBP15- 20 mg/kg 14 Day MAD: Subjects were orally administered VBP15 at 20.0 mg/kg daily for 14 days under fasted conditions.
- Placebo MAD: Subjects were orally administered placebo daily for 14 days under fasted conditions.
Period: Overall Study
Arm/Group | VBP15- 0.1 mg/kg SAD | VBP15- 0.3 mg/kg SAD | VBP15- 1.0 mg/kg SAD | VBP15- 3.0 mg/kg SAD | VBP15- 8.0 mg/kg Fasted SAD | VBP15- 8.0 mg/kg Fed SAD | VBP15- 20.0 mg/kg SAD | Placebo SAD | VBP15- 1.0 mg/kg 14 Day MAD | VBP15- 3.0 mg/kg 14 Day MAD | VBP15- 9.0 mg/kg 14 Day MAD | VBP15- 20 mg/kg 14 Day MAD | Placebo MAD
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 5 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- VBP15- 1.0 mg/kg 14 Days MAD: Subjects were orally administered VBP15 at 1.0 mg/kg daily for 14 days under fasted conditions
- VBP15 - 3.0 mg/kg 14 Days MAD: Subjects were orally administered VBP15 at 3.0 mg/kg daily for 14 days under fasted conditions
- VBP15- 9.0 mg/kg 14 Days MAD: Subjects were orally administered VBP15 at 9.0 mg/kg daily for 14 days under fasted conditions
- VBP15- 20.0 mg/kg 14 Days MAD: Subjects were orally administered VBP15 at 20.0 mg/kg daily for 14 days under fasted conditions
- Total: Total of all reporting groups
Arm/Group | VBP15- 0.1 mg/kg SAD | VBP15- 0.3 mg/kg SAD | VBP15- 1.0 mg/kg SAD | VBP15- 3.0 mg/kg SAD | VBP15- 8.0 mg/kg Fasted SAD | VBP15- 8.0 mg/kg Fed SAD | VBP15- 20.0 mg/kg SAD | Placebo SAD | VBP15- 1.0 mg/kg 14 Days MAD | VBP15 - 3.0 mg/kg 14 Days MAD | VBP15- 9.0 mg/kg 14 Days MAD | VBP15- 20.0 mg/kg 14 Days MAD | Placebo MAD | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8 | 86
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8 | 86
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12 | 6 | 6 | 6 | 6 | 8 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Effects After a Single Dose of VBP15
Time Frame: Participants will be followed for the duration of hospital stay of 4 days
Measure: Number; unit: participants
Groups:
- VBP15- 0.1 mg/kg SAD: Subjects were administered single dose of VBP15 at 0.1 mg/kg under fasted conditions.
- VBP15- 0.3 mg/kg SAD; VBP15- 20.0 mg/kg SAD: Subjects were administered a single dose of VBP15 at 0.3 mg/kg under fasted conditions.
- VBP15- 1.0 mg/kg SAD: Subjects were administered a single dose of VBP15 at 1.0 mg/kg under fasted conditions.
- VBP15- 3.0 mg/kg SAD: Subjects were administered a single dose of VBP15 at 3.0 mg/kg under fasted conditions.
- VBP15- 8.0 mg/kg Fasting SAD: Subjects were administered a single dose of VBP15 at 8.0 mg/kg under fasted conditions.
- VBP15- 8.0 mg/kg Fed SAD: Subjects were administered a single dose of VBP15 at 8.0 mg/kg within 30 minutes of beginning a high-fat/high calorie meal.
- Placebo SAD: Subjects were administered a single dose of placebo under fasted conditions.
Arm/Group | VBP15- 0.1 mg/kg SAD | VBP15- 0.3 mg/kg SAD | VBP15- 1.0 mg/kg SAD | VBP15- 3.0 mg/kg SAD | VBP15- 8.0 mg/kg Fasting SAD | VBP15- 8.0 mg/kg Fed SAD | VBP15- 20.0 mg/kg SAD | Placebo SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12
participants | 2 | 1 | 1 | 1 | 0 | 1 | 0 | 0

2. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) After a Single Dose of VBP15 (0 Through 72 Hours Post Dose)
Time Frame: Participants will be followed for the duration of hospital stay of 4 days
Measure: Mean (Standard Deviation); unit: (hr*ng/mL)
Groups:
- VBP15- 0.1 mg/kg SAD: Subjects were administered a single dose of VBP15 at 0.1 mg/kg under fasted conditions.
- VBP15- 8.0 mg/kg Fasted SAD: Subjects were administered a single dose of VBP15 at 8.0 mg/kg under fasted conditions.
Arm/Group | VBP15- 0.1 mg/kg SAD | VBP15- 0.3 mg/kg SAD | VBP15- 1.0 mg/kg SAD | VBP15- 3.0 mg/kg SAD | VBP15- 8.0 mg/kg Fasted SAD | VBP15- 8.0 mg/kg Fed SAD | VBP15- 20.0 mg/kg SAD | Placebo SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12
(hr*ng/mL) | 42 (17) | 161 (16) | 486 (20) | 1578 (21) | 3997 (55) | 10139 (25) | 8545 (30) | 0 (0)

3. Primary Outcome: Peak Plasma Concentration (Cmax) of VBP15 After a Single Dose of VBP15
Time Frame: Participants will be followed for the duration of hospital stay of 4 days
Measure: Mean (Standard Deviation); unit: (ng/mL)
Arm/Group | VBP15- 0.1 mg/kg SAD | VBP15- 0.3 mg/kg SAD | VBP15- 1.0 mg/kg SAD | VBP15- 3.0 mg/kg SAD | VBP15- 8.0 mg/kg Fasting SAD | VBP15- 8.0 mg/kg Fed SAD | VBP15- 20.0 mg/kg SAD | Placebo SAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 12
(ng/mL) | 13 (13) | 51 (17) | 122 (33) | 305 (24) | 718 (43) | 1817 (31) | 1648 (17) | 0 (0)

4. Primary Outcome: Number of Subjects With Adverse Effects After 14 Daily Doses of VBP15
Time Frame: Participants will be followed for the duration of hospital stay of 15 days
Measure: Number; unit: participants
Groups:
- VBP15- 3.0 mg/kg 14 Days MAD: Subjects were orally administered VBP15 at 3.0 mg/kg daily for 14 days under fasted conditions.
- Placebo MAD: Subjects were orally admistered placebo daily for 14 days under fasted conditions.
Arm/Group | VBP15- 1.0 mg/kg 14 Days MAD | VBP15- 3.0 mg/kg 14 Days MAD | VBP15- 9.0 mg/kg 14 Days MAD | VBP15- 20.0 mg/kg 14 Days MAD | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
participants | 2 | 0 | 0 | 2 | 2

5. Primary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) After 14 Daily Doses of VBP15 (0 Through 72 Hours Post Dose)
Time Frame: Participants will be followed for the duration of hospital stay of 15 days
Measure: Mean (Standard Deviation); unit: (hr*ng/mL)
Arm/Group | VBP15- 1.0 mg/kg 14 Days MAD | VBP15- 3.0 mg/kg 14 Days MAD | VBP15- 9.0 mg/kg 14 Days MAD | VBP15- 20.0 mg/kg 14 Days MAD | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 12
(hr*ng/mL) | 794 (22) | 1494 (19) | 4366 (20) | 9309 (39) | 0 (0)

6. Primary Outcome: Peak Plasma Concentration (Cmax) of VBP15 After 14 Daily Doses of VBP15
Time Frame: Participants will be followed for the duration of hospital stay of 15 days
Measure: Mean (Standard Deviation); unit: (ng/mL)
Arm/Group | VBP15- 1.0 mg/kg 14 Days MAD | VBP15- 3.0 mg/kg 14 Days MAD | VBP15- 9.0 mg/kg 14 Days MAD | VBP15- 20.0 mg/kg 14 Days MAD | Placebo MAD
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 8
(ng/mL) | 153 (16) | 281 (37) | 1082 (23) | 2416 (51) | 0 (0)

ADVERSE EVENTS:
Groups:
- VBP15- 8.0 mg/kg Fed SAD: Subjects were orally administered a single dose of VBP15 at 8.0 mg/kg within 30 minutes of beginning a high-fat/high calorie meal.
- VBP15- 20.0 mg/kg SAD: Subjects were orally administered a single dose of VBP15 at 0.3 mg/kg under fasted conditions.
- VBP15- 1.0 mg/kg 14 Days MAD: Subjects were orally administered a dose of VBP15 at 1.0 mg/kg daily for 14 days under fasted conditions.
- VBP15- 3.0 mg/kg 14 Days MAD: Subjects were orally administered a dose of VBP15 at 3.0 mg/kg daily for 14 days under fasted conditions.
- VBP15- 9.0 mg/kg 14 Days MAD: Subjects were orally administered a dose of VBP15 at 9.0 mg/kg daily for 14 days under fasted conditions.
- VBP15- 20.0 mg/kg 14 Days MAD: Subjects were orally administered a dose of VBP15 at 20.0 mg/kg daily for 14 days under fasted conditions.
- Placebo MAD: Subjects were orally administered a dose of placebo daily for 14 days under fasted conditions.
Arm/Group | VBP15- 0.1 mg/kg SAD | VBP15- 0.3 mg/kg SAD | VBP15- 1.0 mg/kg SAD | VBP15- 3.0 mg/kg SAD | VBP15- 8.0 mg/kg Fasted SAD | VBP15- 8.0 mg/kg Fed SAD | VBP15- 20.0 mg/kg SAD | Placebo SAD | VBP15- 1.0 mg/kg 14 Days MAD | VBP15- 3.0 mg/kg 14 Days MAD | VBP15- 9.0 mg/kg 14 Days MAD | VBP15- 20.0 mg/kg 14 Days MAD | Placebo MAD
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/12 | 0/6 | 0/6 | 0/6 | 0/6 | 0/8
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6 | 1/6 | 1/6 | 0/6 | 1/6 | 0/6 | 0/12 | 2/6 | 0/6 | 0/6 | 2/6 | 2/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VBP15- 0.1 mg/kg SAD (N=6) | VBP15- 0.3 mg/kg SAD (N=6) | VBP15- 1.0 mg/kg SAD (N=6) | VBP15- 3.0 mg/kg SAD (N=6) | VBP15- 8.0 mg/kg Fasted SAD (N=6) | VBP15- 8.0 mg/kg Fed SAD (N=6) | VBP15- 20.0 mg/kg SAD (N=6) | Placebo SAD (N=12) | VBP15- 1.0 mg/kg 14 Days MAD (N=6) | VBP15- 3.0 mg/kg 14 Days MAD (N=6) | VBP15- 9.0 mg/kg 14 Days MAD (N=6) | VBP15- 20.0 mg/kg 14 Days MAD (N=6) | Placebo MAD (N=8)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear Pain, Left (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin, increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain extremity left elbow (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Arthralgia
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Elevated liver enzymes (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Worsening of toothache-right upper molar (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Toothache
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Elevated liver enzyme: ALT (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days